CLINICAL TRIAL: NCT04958551
Title: Basic Research Projects Related to Sports Injuries Such as Degenerative Osteoarthritis, Cruciate Ligament Injury, Patella Dislocation, Discoid Meniscus
Brief Title: Basic Research Projects Related to Sports Injuries
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00006761-M2021180
Record Dates: First submitted 2021-06-24; First posted 2021-07-12 (Actual); Last update posted 2023-06-23 (Actual); Status verified 2023-01

CONDITIONS: Osteoarthritis, Knee; Cruciate Ligament Injury; Patella Dislocation; Discoid Meniscus of Knee
MeSH Terms: conditions — Osteoarthritis, Knee; Patellar Dislocation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, tissue
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
Biological samples are important human genetic resources, which can provide great value for medical research, and how to protect and rationally utilize them is of great importance.However, at present, the blood samples after laboratory examination and the damaged tissue cleaned up in the operation will be treated as medical waste and treated according to the standard of medical waste.However, if these samples can be effectively collected and reasonably used, they can provide extremely high value for the study of sports injury-related diseases.Sports injury and joint structure belongs to multiple factors cause abnormal, through the degenerative osteoarthritis, cruciate ligament injury, patellar dislocation, discoid meniscus injury related basic research project establishment and collect the founding the research institute of sports medicine treated patients with sports injury, including degenerative osteoarthritis, intraoperative tissue, blood and saliva samples,To sample from the micro level of susceptibility genes and molecular signaling pathways to anatomical morphology and histopathologic study direction, and so on, can also for multiple transverse comparison research between samples, in order to investigate sports injury, including degenerative osteoarthritis pathogenesis, for sports trauma related disease etiology, diagnosis, treatment to provide new ideas and methods,And the selection of athletes, athletes special training plans, sports mode to provide more targeted suggestions.This study strictly complied with the Regulations of the People's Republic of China on the Management of Human Genetic Resources to establish the Institute of Sports Medicine Sample Bank, which can reduce the waste of human genetic resources in China, promote the development of the discipline, and provide a higher platform for the study of sports injure-related diseases.

DETAILED DESCRIPTION:
I. Research Background In the "Twelfth Five-Year Plan for Biotechnology Development", the requirements for the construction of national biological science facilities are clearly put forward, and the construction of a national biological center, which includes the biological technology management information database and biological sample resource database.Biobank mainly refers to the standardized collection, processing, storage and application of biomacromolecules, cells, tissues and organs of healthy and disease organisms, including human organ tissues, whole blood, plasma, serum, biological fluid or processed biological samples (DNA, RNA, protein, etc.).Establish a standardized quality control, information management and application system for samples 1.In 1987 the American Institute of Cancer Research established a biobank of cancer samples.The UK Biobank was set up in 1999 to collect and closely monitor samples from 500,000 volunteers.At the same time, domestic and foreign research institutions are also jointly building and sharing biobanks.Europe, for example, has carried out genetic studies involving 520,000 people in 23 sample centers in 10 European countries.Human genetic resources are important strategic resources, China has a unique advantage of human genetic resources, effective protection and rational use of human genetic resources is very important.Proper collection of abundant and large sample resources is bound to provide great value for biological and medical research 3.

Sports medicine institute, Peking University third hospital is the largest sports medicine center, about 120000 m years MenZhenLiang, nearly 10000 years since, before the operation exsanguinate assay blood samples in laboratory tests, after the completion of the operation clean up the damage of tissue samples at the end of the surgery, for medical waste, by medical waste treatment, but the samples has high research value.From including morphological, genetic and molecular mechanism study 4-6, for sample tissue pathological slices, gene sequencing and other research methods to the field of sports medicine related diseases have a deeper understanding, and provide samples for future researchers reserve platform, to build samples of sports medicine institute library.

Sports injuries and joint structural abnormalities are multi-factor causes. Through the establishment of this project and the collection of intraoperative tissue, blood and saliva samples from patients with sports injuries, including degenerative osteoarthritis, admitted to the Institute of Sports Medicine of the Third Hospital of Beijing Medical University,To sample from the micro level of susceptibility genes and molecular signaling pathways to anatomical morphology and histopathologic study direction, and so on, can also for multiple transverse comparison research between samples, in order to investigate sports injury, including degenerative osteoarthritis pathogenesis, for sports trauma related disease etiology, diagnosis, treatment to provide new ideas and methods,And the selection of athletes, athletes special training plans, sports mode to provide more targeted suggestions.

II. Research Objectives

1. After the completion of the laboratory examination, the blood samples and tissue samples and body fluids discarded during the operation are retained for the purpose of building the "Basic Research Project on Sports Injuries Related to Degenerative Osteoarthritis, Cruciate Ligament Injury, Patella Dislocation, Discoid Meniscus and so on".
2. Use the samples of "Basic Research Project on Sports Injury Related to Degenerative Oosteoarthritis, Cruciate Ligament Injury, Patella Dislocation, Discoid Meniscus and Other Sports Injury" to conduct related research on the mechanism of sports injury, new treatment methods and treatment techniques to improve the efficacy.

III. Experimental design:

1. Biological sample collection 1.1 Target population of sample collection Outpatients, inpatients, follow-up patients and third-class blood relatives or close relatives of patients with degenerative osteoarthritis, cruciate ligament injury, patella dislocation, discoid meniscus who were admitted to the Institute of Sports Medicine of the Third Hospital of Peking University voluntarily enrolled in the biobase.

1.2 Sample collection and preservation

1. For patients undergoing sports injury surgery, intraoperative tissue stump (divided into 2 pieces) and remaining whole blood samples (1.5 mL/piece, a total of 3 pieces) were mainly collected. Meanwhile, genetic information was extracted and preserved for some samples.In strict accordance with the standardized operation process of project samples, samples are processed and stored separately in the warehouse, and stored in the -80℃ ultra-low temperature refrigerator or -196℃ liquid nitrogen tank.Patient related imaging and surgical data were recorded and saved by the hospital system.
2. The remaining whole blood samples (1.5 mL/piece, 3 pieces in total) and saliva samples (about 3 mL/piece) were mainly collected from the other subjects except the patients undergoing surgery. At the same time, genetic information of some samples was extracted and stored.In strict accordance with the standardized operation process of project samples, samples are processed and stored separately in the warehouse, and stored in the -80℃ ultra-low temperature refrigerator or -196℃ liquid nitrogen tank.Relevant imaging and surgical data were recorded from previous medical records or provided by the subjects themselves.

2. Biobank preservation and management The biobank is in strict compliance with the Regulations of the People's Republic of China on the Management of Human Genetic Resources for sample storage, processing and management.

2.1 Quality control of sample warehousing In strict accordance with the standardized operation process of project samples, samples are processed and stored separately in the warehouse, and stored in the -80℃ ultra-low temperature refrigerator or -196℃ liquid nitrogen tank.For genetic extraction of tissue samples, blood and saliva samples, ensure that the total number of samples is at least 1ug, and ensure that the sample OD 260/280 is close to 2.0.

2.2 Sample information management The sample information was managed electronically by the biobank information management system of Peking University Third Hospital.Keep full operation records including sample processing, packing, warehousing, quality inspection, freeze-thaw, loss reporting, etc., and relevant documents signed by the operator.

2.3 Safety of sample environment The environmental safety of samples is managed according to the standard of the biobank of Peking University Third Hospital. Automatic monitoring system of temperature, humidity and environment is adopted to collect and record the samples in real time.In case of any abnormality, the system will inform the management staff of the biobank of the Institute of Sports Medicine of our hospital through SMS.

2.4 Regular quality inspection of samples Quality tests were carried out according to the standards of the biobank of Peking University Third Hospital. Quality tests of DNA, RNA, tissue samples and cell activity were carried out regularly to ensure the accuracy of the results obtained from the samples for subsequent studies.

3. Basic research related to biological samples The collected biological samples were sequenced and analyzed for genetic information, tissue morphology, and expression determination and analysis of related biomolecules.

Four, data management:

1. Data entry:

   According to the original observation records of the subjects, the researchers will timely, complete, correct and clear data into the case report form.After being reviewed and signed by the principal investigator, the questionnaire should be sent to the clinical study data administrator in a timely manner.
2. Contents and methods of data verification and management:

   When all case report forms are checked without error, the data manager will write the database inspection report, which includes the study completion status (including the list of exclusions), inclusion/exclusion criteria, integrity check, logical consistency check, outlier data check, time window check, adverse event check, etc.

   At the audit meeting, the principal investigator, data administrator and statisticians will make decisions on subjects' signing of informed consent and questions raised in the database inspection report, and write the audit report. The database will be locked at the same time.
3. Data archiving:

After data entry and verification as required, the case report form shall be archived in numbered order and filled in with the retrieval directory for future reference.Electronic data files, including databases, inspection procedures, analysis procedures, analysis results, codebooks and explanatory files, should be classified and stored in multiple backups on different disks or recording media. They should be properly stored to prevent damage.All original files shall be kept for the specified period of time.

V. Safety evaluation:

There is no special risk associated with participation in this study.The sampling process of tissue samples will not affect the quantity and quality of blood tests and examinations of patients before surgery, nor will it affect the surgical method of patients, nor will it affect the choice of surgical method by the surgeon. Therefore, there will be no change in preoperative preparation, intraoperative operation and surgical effect, and there will be no related risks.

Participation in this study will not increase any medical history and illness inquiries, physical examination content, blood tests, auxiliary examinations such as X-ray, CT, MRI and B-mode ultrasound, and will not increase any fees.

VI. Subject Protection (Informed Consent, Subject's Benefits and Risks, Confidentiality, Conflict of Interest and Other Ethical Consideration) According to relevant Chinese laws and regulations, before the start of the study, the researcher shall give written and oral explanations to the subjects regarding the background, nature, significance, steps, benefits, risks and withdrawal of the study, etc., and an informed consent signed by each subject (or legal representative of the subject) shall be obtained.The informed consent form is dated and its copy is kept separately by the investigator and the subject.

Seven, research management

1. Scheme modification (define the principle and process of scheme modification after the project starts) It could be that the researchers found persistent non-compliance with the inclusion criteria caused the change, or it could be that the inclusion criteria were too strict and the number of recruits was too low.Revision of changes in this part of the study protocol should take into account any statistical effects, such as adjustment of sample size due to changes in event rates, or revision of the analysis plan.
2. Quality management (project supervision plan) :

Specific monitoring contents include:

1. The verification scheme shall be submitted to the ethics committee for approval.
2. The researchers participating in this validation conscientiously followed the standard operating procedures for clinical validation before, during and after the validation.
3. During the verification process, the researcher monitored the correctness and integrity of the data in CRF.
4. According to the requirements of the case report form, researchers should faithfully, carefully and carefully record all contents in CRF to ensure that the contents of the case report form are true and reliable.
5. All observations and findings in clinical validation should be verified to ensure the reliability of data, ensure that all conclusions in clinical validation are derived from original data, and appropriate data management measures should be taken in clinical validation and data processing.

3. Early Termination:

Define the principles and treatment for early termination of study, such as:

If serious adverse reactions occur in the trial, the clinical trial should be terminated in time.

Serious deviations were found in the implementation of clinical trials and it was difficult to evaluate the efficacy of surgical treatment.

The applicant requests termination or the administration requests termination of the experiment.

ELIGIBILITY:
Inclusion criteria:

1. Outpatients, inpatients, follow-up patients and third-class blood relatives or close relatives of patients with degenerative osteoarthritis who were admitted to the Institute of Sports Medicine of the Third Hospital of Peking University, the Second Affiliated Hospital of Xinjiang Medical University，and Hebei Cangzhou Hospital of Integrated Traditional Chinese and Western Medicine voluntarily enrolled in the biobase.
2. Outpatients, inpatients, follow-up patients and third-class blood relatives or close relatives of patients with cruciate ligament injury who were admitted to the Institute of Sports Medicine of the Third Hospital of Peking University voluntarily enrolled in the biobase.
3. Outpatients, inpatients, follow-up patients and third-class blood relatives or close relatives of patients with patella dislocation who were admitted to the Institute of Sports Medicine of the Third Hospital of Peking University voluntarily enrolled in the biobase.
4. Outpatients, inpatients, follow-up patients and third-class blood relatives or close relatives of patients with discoid meniscus who were admitted to the Institute of Sports Medicine of the Third Hospital of Peking University voluntarily enrolled in the biobase.

Exclusion criteria: -.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Outpatients, inpatients, follow-up patients and third-class blood relatives or close relatives of patients with degenerative osteoarthritis, cruciate ligament injury, patella dislocation, discoid meniscus who were admitted to the Institute of Sports Medicine of the Third Hospital of Peking University, the Second Affiliated Hospital of Xinjiang Medical University，and Hebei Cangzhou Hospital of Integrated Traditional Chinese and Western Medicine voluntarily enrolled in the biobase.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2021-04-10 (Actual); Primary Completion 2024-07-30 (Estimated); Study Completion 2025-07-10 (Estimated)

PRIMARY OUTCOMES:
DNA-seq | up to 2 weeks
  Whole genome sequencing
Clinical information collection | up to 2 weeks
  basic information, radiological measurements and physical examination

CONTACTS AND LOCATIONS:
Overall Officials: Jia-kuo Yu, Phd., Study Chair — Institute of Sports Medicine, Peking University Third Hospital, Beijing, China, 100191
Locations (1):
- Institute of Sports Medicine, Peking University Third Hospital, Beijing, Beijing Municipality, China